CLINICAL TRIAL: NCT04412031
Title: Bayesian Network to Predict Transfer in Intensive Care Units or Death in Newly Covid-19 Hospitalized Patient
Brief Title: Prediction of Unfavourable Outcome in Newly Covid-19 Hospitalized Patient
Acronym: PredictCovid19
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 20_185
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: to Predict an Unfavorable Evolution of Covid-19 at the Hospital Admission of Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non applicable — non applicable

SUMMARY:
The project is a part of the "Protocol for a multicentre study of nosocomial SARS-CoV2 transmission: The NOSO-COR Project" registered in ClinicalTrials (NCT04290780).

In the current pandemic context, medical resources have often been exceeded. Developing, using artificial intelligence techniques, an algorithm capable of detecting patients at risk of acute respiratory distress following Sars-Cov2 infection could help physicians to optimize the treatment of patients and health decision-makers to optimize resources. Thus, the goal of this project is to create a prediction model using artificial intelligence to predict an unfavorable evolution of Covid-19 at the hospital admission of patients

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years or older at the time of signing the informed consent
* Volunteer patients, care givers and healthcare professionals in France and hospitals affiliated with the GABRIEL network. Demographic and clinical data will be collected using case-report forms designed especially for the purpose of the project.
* A nasopharyngeal swab will be collected and tested for SARS-CoV2 by RT-PCR.
* Admission to hospital

Exclusion Criteria:

* Age lower than 18 years old
* Patients protected by the law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The project is a part of the "Protocol for a multicentre study of nosocomial SARS-CoV2 transmission: The NOSO-COR Project"
  It is an international multicentre prospective, observational, hospital-based study in adults. It will include volunteer patients, care givers and healthcare professionals in France and hospitals affiliated with the GABRIEL network. Demographic and clinical data will be collected using case-report forms designed especially for the purpose of the project. A nasopharyngeal swab will be collected and tested for SARS-CoV2 by RT-PCR. Characteristics of the study participants, the proportion of confirmed nosocomial SARS-CoV2 infections relative to all patients with syndromes suggestive of 2019-nCoV infection will be analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 802 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Need of mechanical ventilation, transfer to an intensive care unit or death within 21 days of admission. | within 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital E Herriot - Hospices Civils de LYON, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided